CLINICAL TRIAL: NCT01687465
Title: A Randomized Clinical Trial of Selective Laser Trabeculoplasty (SLT) in Open Angle Glaucoma Who Had Been Previously Treated With Complete SLT
Brief Title: A Trial to Compare the Laser Treatment (SLT vs. ALT) in Glaucoma Patients
Acronym: SLTRepeat
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, William Hodge, Professor of Department of Ophthalmology, Western University, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR granted glaucoma RCT
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
Keywords: glaucoma; laser; SLT; ALT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argon laser trabeculoplasty (Active Comparator): Up to the year 2005, the vast majority of ophthalmologists used Argon laser trabeculoplasty (ALT) as the mode of laser therapy. ALT is effective but its most significant problem is that its effectiveness decreases with re-treatment since the tissue it targets (the trabecular meshwork) is changed by the laser rendering repeat treatments less effective.
  Interventions: Procedure: Argon laser trabeculoplasty; Procedure: Selective laser trabeculoplasty
- selective laser trabeculoplasty (Active Comparator): Post 2005, a newer mode of laser therapy, selective laser trabeculoplasty (SLT) has emerged as the standard of care laser. There are many potential advantages to SLT but to date these advantages are only theoretical. The most important potential clinical advantage of SLT is that it causes less damage to the tissue it targets.
  Interventions: Procedure: Argon laser trabeculoplasty; Procedure: Selective laser trabeculoplasty

INTERVENTIONS:
Procedure: Argon laser trabeculoplasty — With Argon laser trabeculoplasty (ALT), thermal energy is used directed towards the Trabecular Meshwork (the site of aqueous drainage from the eye),which causes focal scarring of trabecular meshwork, thus enable fluid drainage more effectively. However, this procedure may not be repeatable since it causes too much damage to the trabecular meshwork.
Procedure: Selective laser trabeculoplasty — Selective laser trabeculoplasty is a relatively newer technology that uses a Nd:YAG laser to target specific cells within the trabecular meshwork. SLT does not cause coagulative damage to the trabecular meshwork, and thus has the advantage of being repeatable.

SUMMARY:
Lasers are important therapy in glaucoma. They are a pivotal point in treatment between medical and surgical care. Over the last 10 years a new laser has emerged as the usual laser treatment: Selective laser trabeculoplasty (SLT). SLT works as well as the older laser used: argon laser trabeculoplasty (ALT). However SLT has many theoretical benefits over ALT including causing less damage to the tissue it affects. One of the potential patient centered benefits of this laser is that it may be repeatable. It is even possible that the old laser ALT may be useable after an SLT treatment. This study aims to uncover whether repeat laser is possible after SLT and if so which laser is more effective (ALT vs SLT). The potential of repeating laser therapies may delay surgical treatment and its complications. Also understanding which laser to use will help eye doctors know how to treat their patients at this point of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Over age of 18 yo.
* OAG including pigmentary dispersion syndrome and pseudoexfoliation
* OAG has been treated with 360 degrees of SLT
* two sighted eyes,
* willing to participate after being informed of and reading the patient information material.

Exclusion Criteria:

* Narrow angle glaucoma
* Previous glaucoma surgery
* Eye surgery expected in the next 12 months
* Severe corneal disease
* On or anticipated steroid in 6 months
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 12 months post operatively
  IOP difference between baseline and 12 month post-laser.

SECONDARY OUTCOMES:
To compare the IOP lowering effect between the groups at other postoperative visits | 12 months
  IOP difference between baseline, 1hr, 1 wk, and 1, 3, 6 and 12 mon post-laser.
To compare the visual acuity between the groups at all visits. | 12 months
  VA difference between baseline, 1hr, 1 wk, and 1, 3, 6 and 12 mon post-laser.
To compare the trabecular meshwork pigmentation between the groups at all visits. | 12 months
To compare any adverse events between the two groups at all visits. | 12 months
SLT repeatability of long term follow up in glaucoma patients | 36 months after initial enrollment of the primary study
  The follow up time has been extended two more years. Patients will be followed up Q6 months.

CONTACTS AND LOCATIONS:
Overall Officials: William G Hodge, MD, PhD, Principal Investigator — Lawson Research Institute, Univ. of Western Ontario
Locations (7):
- Canada (7):
  - Rockyview General Hospital, University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, University of Alberta, Edmonton, Alberta
  - Eye Care Centre, Dalhousie University, Halifax, Nova Scotia
  - McMaser University, St. Joseph's Healthcare Hamilton, CAHS Regional Eye Institute, Hamilton, Ontario
  - Ivey Eye Institute, St. Joseph's Hospital, Western University, London, Ontario
  - Sunnybrook Health Sciences Centre, University of Toronto, Toronto, Ontario
  - McGill University, Dept. of Ophthalmology, Royal Victoria Hospital,, Montreal, Quebec

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114
- [Derived] Hutnik C, Crichton A, Ford B, Nicolela M, Shuba L, Birt C, Sogbesan E, Damji KF, Dorey M, Saheb H, Klar N, Guo H, Hodge W. Selective Laser Trabeculoplasty versus Argon Laser Trabeculoplasty in Glaucoma Patients Treated Previously with 360 degrees Selective Laser Trabeculoplasty: A Randomized, Single-Blind, Equivalence Clinical Trial. Ophthalmology. 2019 Feb;126(2):223-232. doi: 10.1016/j.ophtha.2018.09.037. Epub 2018 Sep 29. PMID 30278197